CLINICAL TRIAL: NCT05816798
Title: Photobiomodulation in Chronic Knee Pain in Patients Who Are in PreRehabilitation for Bariatric Surgery: Double Blind, Randomized, Controlled Placebo Clinical Trial
Brief Title: Photobiomodulation in Chronic Knee Pain in Patients Who Are in PreRehabilitation for Bariatric Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Rebeca Boltes Cecatto, MD., PhD. Researcher, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhotobioKneepain
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Knee Pain; Obesity, Morbid
Keywords: Photobiomodulation; Chronic knee pain; Obesity Morbid; Central and periferic sensitivity; Nociception
MeSH Terms: conditions — Obesity, Morbid | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant: The participant will be blind to the group they will be participating in. The device display will be hidden so the patient cannot see if it is on or off. The device activation noise will be recorded and used to mimic the irradiation.
  Principal Investigator: only the auxiliary investigator who will apply the laser will know the group of participants. The principal investigator performing the initial and final (post-treatment) assessments will be blinded to the treatment/placebo groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation Intervention (Experimental): PBM therapy sessions will be performed with the Therapy EC device (DMC brand) 100mW power, which is a Low Intensity Laser Therapy. During the interventions, the patient will be allowed to choose the position that is most comfortable for him and accompanied by the physical therapist throughout the procedure. Examiner and patient will be wearing protective eyewear. Applications will occur after local asepsis of the device and skin. Patients will receive the PBM therapy described below:
  * Paravertebral region at levels L3 to S2:1 cm lateral to the corresponding level, on each right and left side, which are root levels that innervate the knee joint (totaling 10 paravertebral points) with 3 Joules per point (30 s) in each point
  * Knees bilaterally (4 points each knee): anteromedial portal; anterolateral portal; apex of patella; base of patella; with 4 J per point (40 s)
  Interventions: Device: Photobiomodulation; Other: Standard Physiotherapy Tretament
- Photobiomodulation Placebo (Placebo Comparator): Control group research participants will receive the standard treatment described as well as placebo PBM treatment to mask the treatment. The number of points, dose and PBM application site will be the same as described in the PBM Intervention Group item, however the PBM equipment will be turned off.
  Interventions: Other: Standard Physiotherapy Tretament; Device: Photobiomodulation Placebo

INTERVENTIONS:
Device: Photobiomodulation — PBM is a therapeutic technique that uses light at different wavelengths (red or infrared), in a non-invasive way in which non-ionizing irradiation is used to produce a series of photophysical and photochemical effects when applied to biological tissues (humans and animals). Regarding the clinical results, numerous articles have already demonstrated the effect of PBM in improving pain and disability in patients with knee joint pain.
  Other Names: Low level laser therapy
  Arms: Photobiomodulation Intervention
Other: Standard Physiotherapy Tretament — standard treatment (physiotherapy-standard exercises: Cardiopulmonary physiotherapy and Physiotherapy with global muscle strengthening exercises). This program will be maintained for all study patients, for both groups, throughout the data collection period and includes activities 2X per week.)
Device: Photobiomodulation Placebo — The same interventions described of Photobiomodulation Group bu device will be turned off
  Arms: Photobiomodulation Placebo

SUMMARY:
Chronic pain is a global public health problem, which intensifies even more in the obese population, reaching about 33% of these patients. Among the topography, chronic knee pain affects 80%, constituting an important cause of disability and decreased quality of life. In addition, in grade 3 obesity, also called morbid obesity, in which bariatric surgery is already indicated, knee pain makes it difficult or prevents participation in the pre-habilitation program that includes physical therapy through therapeutic exercises with the aim of reducing postoperative complications. In this sense, a double-blind, randomized, placebo-controlled clinical trial will be conducted with the objective of evaluating the effect of photobiomodulation (PBM) on pain and functionality of obese patients with chronic knee pain who are in a prehabilitation program for bariatric surgery, discussing its role as an analgesic therapy and modifier of peripheral and central sensitization mechanisms of the pain pathway. PBM is a safe treatment option, with no undesirable effects and low cost. The primary outcomes will be pain intensity, through visual analogue scale, and Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire, validated version for Portuguese - Brazil. Secondary outcomes will be pressure pain threshold and rolling pinch maneuver measured by digital algometer. Other exploratory outcomes will be 6-minute walk test, knee range of motion, SF-36 quality of life questionnaire. There will be 2 groups: an intervention group (photobiomodulation associated with standard physiotherapy treatment) and another placebo group (device turned off associated with the same standard physiotherapy treatment). The application sites will be knees and lumbar paravertebral 2 times a week for 12 weeks. The dosimetric standards will be 4J/point in the knees and 3J/point in the lumbar. The results obtained will be statistically analyzed and later published in a scientific journal.

DETAILED DESCRIPTION:
Chronic pain is a global public health problem, which intensifies even more in the obese population, reaching about 33% of these patients. Among the topography, chronic knee pain affects 80%, constituting an important cause of disability and decreased quality of life. In addition, in grade 3 obesity, also called morbid obesity, in which bariatric surgery is already indicated, knee pain makes it difficult or prevents participation in the pre-habilitation program that includes physical therapy through therapeutic exercises with the aim of reducing postoperative complications. In this sense, a double-blind, randomized, placebo-controlled clinical trial will be conducted with the objective of evaluating the effect of photobiomodulation (PBM) on pain and functionality of obese patients with chronic knee pain who are in a prehabilitation program for bariatric surgery, discussing its role as an analgesic therapy and modifier of peripheral and central sensitization mechanisms of the pain pathway. PBM is a safe treatment option, with no undesirable effects and low cost. The primary outcomes will be pain intensity, through visual analogue scale, and Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire, validated version for Portuguese - Brazil. Secondary outcomes will be pressure pain threshold and rolling pinch maneuver measured by digital algometer. Other exploratory outcomes will be 6-minute walk test, knee range of motion, SF-36 quality of life questionnaire. There will be 2 groups: an intervention group (photobiomodulation using Therapy EC-DMC device associated with standard physiotherapy treatment) and another placebo group (device turned off associated with the same standard physiotherapy treatment). The application sites will be knees (4 anatomically described points) and lumbar paravertebral (levels L3 to S2 bilateral - 10 points, being 05 points each side) 2 times a week for 12 weeks. The dosimetric standards will be 4J/point (40 seconds) in the knees and 3J/point (30 seconds) in the lumbar. The results obtained will be statistically analyzed using SPSS 28.0 software, and later published in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with indication for bariatric surgery performed in routine follow-up at the Gastric Surgery Outpatient Clinic of HC-UFG;
* Patients with chronic pain (> 3 months) in the knees bilaterally. Patients will be asked in the initial evaluation if they feel pain located in the topography of the knees that has been compromising their functionality both in daily activities and at work, and that lasts for more than or equal to 3 months. This pain may be reported as continuous or intermittent;
* Sign the Informed Consent Term approved by the HC-UFG Ethics Committee.

Exclusion Criteria:

* - Loss of follow-up in the outpatient clinic of origin and in the Physiotherapy sector, even though the use of laser therapy was maintained according to the study protocol;
* Any reported adverse effects from the use of FBM reported;
* Patients in whom there are changes in the medications being used for chronic pain during the study protocol will be excluded from this study. Minimal changes in the dosages of medications already in use can be tolerated, as long as there are no changes in the type of medication, but only in the prescribed dose. These modifications throughout the study, if they occur, will be described.
* Death
* Withdrawal of the informed consent by the participant
* If the patient, for any reason, is excluded from the indication of bariatric surgery
* Emergence during the study of any of the non-inclusion criteria, like: .
* Patients with other rheumatologic diseases and/or systemic inflammatory diseases (rheumatoid arthritis, Reiter's arthritis, ankylosing spondylitis, generalized polyarthritis) or previous musculoskeletal diseases in the knees;
* Clinical manifestations or complaints of knee arthralgia related to diseases other than obesity.
* Previous use in the last 90 days of treatment with the use of Phototherapy for the same or another indication;
* Clinical signs of neuropathy, including radiculopathies and peripheral nerve injuries;
* Pain in the lower limb, originating from the lumbar spine (lombosciatalgia)
* Use of corticosteroids at an immunosuppressive dose (20mg daily of prednisone or equivalent for at least 14 days);
* Infection or tumor at the site of therapy application;
* Current chronic infections such as tuberculosis or chronic hepatitis treated or not.
* Blood clotting disorders (including thrombosis) at the application site.
* Diagnosis of fibromyalgia;
* Serious psychiatric disorders that require psychiatric care;
* Systemic injections and/or joint injections of corticosteroids or hyaluronic acid during the last 48 hours prior to the initial assessment of the study;
* Psychoaffective disorder that compromises adherence to treatment;
* Any history of sensitivity to light or phototherapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  10 cm ruler with Visual Analog Pain Scale where 0 indicates no pain and 10 indicates maximum pain possible
Knee injury and Osteoarthritis Outcome Score (KOOS) Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  A specific scale for patients with knee pain

SECONDARY OUTCOMES:
The dermatomes pinching and rolling maneuver Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  The pinching and rolling maneuver in the L1, L2, L3, L4, L5, S1 and S2 dermatomes will also be performed to assess signs of subcutaneous hyperalgesia and the pain threshold will be measured with an algometer.
Pressure pain thresholds will be assessed in the muscles related to knee Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  Pressure pain thresholds will be evaluated with algometer in the muscles: vastus medialis, adductor longus, rectus femoris, vastus lateralis, tibialis anterior, peroneus longus, popliteus, sartorius, gracilis, quadratus lumborum, supraspinatus ligaments (Lumbar) between L1-L2, L2- L3, L3-L4, L4-L5 and L5-S1 and sacral (S) S1-S2, as previously described in the literature

OTHER OUTCOMES:
6 minute walk test Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  This is a routine test on the service to assess functionality
Short Form Health Survey 36 (SF-36) Scale Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  Scale that assesses quality of life and it presents a score that ranges from 0 (zero) to 100 (obtained through Raw Scale calculation), where zero corresponds to the worst general state of health and 100 corresponds to the best state of health
Knee joint range of motion Change | At the initial assessment (baseline in the same day of first PBM therapy) and at the end of the intervention (after 14 weeks from baseline)
  It will be measured with goniometer. Patients will be placed in a sitting position with the trunk supported on the chair, and they will be asked to extend the knee. The fulcrum of the goniometer will be next to the lateral condyle of the femur, one arm will be in line with the lateral malleolus and the other in line with the greater trochanter. And the measure of the angle in the maximum range of motion will be the outcome to be compared.
Preliminary pilot statistical analysis | May 2025
  In an initial pilot evaluation checking safety trends, initial efficacy, or need for sample size adjustments, data from the first 23 participants that complete the intervention protocol, will be statistically analyzed (9 from PBM group and 11 from placebo group).

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca B Cecatto, MD PHD, Principal Investigator — Nove de Julho University
Locations (1):
- Gastric Outpatient Clinic of HC-UFG, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The plan of Data Manage are available in
  https://doi.org/10.48321/D1MW8J Rebeca Cecatto. (2023). "Photobiomodulation in Chronic Knee Pain in Patients Who Are in PreRehabilitation for Bariatric Surgery: Double Blind, Randomized, Controlled Placebo Clinical Trial " [Data Management Plan]. DMPTool. https://doi.org/10.48321/D1MW8J
Supporting Information: Study Protocol, CSR
Time Frame: The registered study protocol will be submitted to publication in a scientific journal making the protocol public before the collected data. Upon completion of the study, the original clinical non-identifiable data referring to pain, quality of life and functionality assessments will be made available in repository, with the purpose of collaborating with the scientific community and auditing. These data collected and stored in the spreadsheets drives will be exported to an Open Science repository such as Mendeley Data, Figshare or similar. The results after the statistical analysis will also be sent for publication in indexed scientific journals.
Access Criteria: follow the policies of these platforms and scientific journals
URL: https://doi.org/10.48321/D1MW8J

REFERENCES:
- [Result] Chen X, Tang H, Lin J, Zeng R. Causal relationships of obesity on musculoskeletal chronic pain: A two-sample Mendelian randomization study. Front Endocrinol (Lausanne). 2022 Aug 23;13:971997. doi: 10.3389/fendo.2022.971997. eCollection 2022. PMID 36082069
- [Result] Chin SH, Huang WL, Akter S, Binks M. Obesity and pain: a systematic review. Int J Obes (Lond). 2020 May;44(5):969-979. doi: 10.1038/s41366-019-0505-y. Epub 2019 Dec 17. PMID 31848456
- [Result] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Result] Hamblin MR. Mechanisms and applications of the anti-inflammatory effects of photobiomodulation. AIMS Biophys. 2017;4(3):337-361. doi: 10.3934/biophy.2017.3.337. Epub 2017 May 19. PMID 28748217
- [Result] Dompe C, Moncrieff L, Matys J, Grzech-Lesniak K, Kocherova I, Bryja A, Bruska M, Dominiak M, Mozdziak P, Skiba THI, Shibli JA, Angelova Volponi A, Kempisty B, Dyszkiewicz-Konwinska M. Photobiomodulation-Underlying Mechanism and Clinical Applications. J Clin Med. 2020 Jun 3;9(6):1724. doi: 10.3390/jcm9061724. PMID 32503238
- [Derived] Amorim ACFG, Belchior TCF, Silva Rodarte TND, Reboucas Junior FA, Rodrigues MFSD, Marcos RL, Lino-Dos-Santos-Franco A, Cecatto RB. Photobiomodulation therapy for chronic knee pain in obese patients in pre-rehabilitation for bariatric surgery: randomised, placebo-controlled, double-blinded, clinical trial protocol. BMJ Open. 2024 Jul 1;14(6):e079864. doi: 10.1136/bmjopen-2023-079864. PMID 38951012